CLINICAL TRIAL: NCT06895226
Title: Exercise and Physical Activity in Adults with Acquired Brain Injury
Acronym: PA_ABI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Andrea Gutiérrez Suárez, PhD, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PA_ABI
Record Dates: First submitted 2025-03-05; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acquired Brain Injury
Keywords: Acquired brain injury; physical activity; intervention
MeSH Terms: conditions — Brain Injuries; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Exercise and physical activity program and usual care (Experimental): Exercise and physical activity program and usual care
  Interventions: Behavioral: Exercise; Other: Usual Care
- Control: usual care (No Intervention): Only usual care

INTERVENTIONS:
Behavioral: Exercise — Exercise and physical activity program and usual care
  Arms: Experimental: Exercise and physical activity program and usual care
Other: Usual Care — Usual cara and Exercise and PA recommendations
  Arms: Experimental: Exercise and physical activity program and usual care

SUMMARY:
Exercise and physical activity in adults with acquired brain injury

DETAILED DESCRIPTION:
Although emerging approaches have emerged in the design of interventions that promote an orientation towards physical activity scientific evidence on their efficacy in this particular population remains limited. This underscores the need for further research to evaluate the efficacy of these intervention approaches in the context of ABI.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years of age and present a medical diagnosis of acquired brain injury.
* Have the informed consent completed and signed
* Present a state that allows following indications for the practice of exercise and physical activity.

Exclusion Criteria:

* Have medical comorbidities that contraindicate the safe performance of the program (i.e., cardiac or respiratory instability, uncontrolled seizures).
* Have additional disabling conditions, such as cognitive impairment and/or an inability to communicate with the researcher verbally, in writing, or through an emissary.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Health-related Quality of Life | Baseline an through study completion, an average of 1 year
  Euroqol 5d Quality of Life outcome
Physical Actvity | Baseline an through study completion, an average of 1 year
  International Physical Actvity Questionnaire